CLINICAL TRIAL: NCT05962463
Title: Comparison of the Effectiveness of Pulsed Radiofrequency Therapy and Canal Adductor Blockade for Chronic Pain and Functioning in Knee Osteoarthritis
Brief Title: Pulsed Radiofrequency Therapy vs Canal Adductor Blockade in Knee Osteoarthritis
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Mensur Salihovic, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: 0120-464/2022/6
Record Dates: First submitted 2023-06-02; First posted 2023-07-27 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
Keywords: Adductor canal blockade; Radiofrequency therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Canal adductor blockade: After surgical cleaning of the anteromedial thigh, all participants in this group received single shot ultrasound guided canal adductor blockade with 14 ml 0,25% levobupivacaine and 100 mcg clonidine mixed in the same syringe. Investigators previously scanned the adductor canal and chose the middle of the canal as the entry point of the 10 cm echogenic ultrasound needle. After the blockade, all participants were monitored in our ambulance for the next hour.
  Interventions: Procedure: Canal adductor blockade
- Pulsed radiofrequency therapy: After surgical cleaning of the anteromedial thigh, all participants in this group received ultrasound-guided pulsed radiofrequency therapy. Investigators previously scanned the adductor canal and chose the middle of the canal as the entry point of the RF 10 cm needle with a 1 cm free tip. After sensory and motor checking all patients have gotten 6 minutes of therapy divided into 3 sequences of 2 minutes of 50 V current and 42. Before starting the PRF therapy all participants have gotten 2 ml 0,25% levobupivacaine through the needle for preventing discomfort during the procedure. After the treatment, all participants were monitored in our ambulance for the next hour.
  Interventions: Procedure: Canal adductor pulsed radio-frequency therapy

INTERVENTIONS:
Procedure: Canal adductor blockade — The same experienced anesthesiologist has performed all blocks. Always after surgical cleaning of the anteromedial thigh, all participants in this group received single shot ultrasound guided canal adductor blockade. After the blockade, all participants were monitored in our ambulance for the next hour.
  Groups: Canal adductor blockade
Procedure: Canal adductor pulsed radio-frequency therapy — The same experienced anesthesiologist has performed all PRF therapy After surgical cleaning of the anteromedial thigh, all participants in this group received ultrasound-guided pulsed radiofrequency therapy. We've previously scanned the adductor canal and chose the middle of the canal as the entry point of the RF 10 cm needle with a 1 cm free tip. After sensory and motor checking all patients have gotten 6 minutes of therapy divided into 3 sequences of 2 minutes of 50 V current and 42ºC. After the treatment, all participants were monitored in our ambulance for the next hour.
  Groups: Pulsed radiofrequency therapy

SUMMARY:
This study is intended to prove the efficacy and safety of ultrasound-guided pulsed radiofrequency therapy on adductor canal nerves by patients with Knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is a serious epidemiologic problem. Non-surgical methods are shown limited efficacy in relieving chronic knee pain in patients in advanced stages of knee osteoarthritis. The knee prosthesis is a successful treatment for many patients with advanced knee osteoarthritis. Still, there are important numbers of patients, which are not appropriate candidates for such surgery treatment or refused surgery for any reason. For them, any treatment which could relieve pain in their knee would have a good impact on their quality of life. Interventions like adductor canal block(ACB) and pulsed radiofrequency therapy (PRF) have demonstrated good results. In this study, investigators compare the effectiveness of these two methods. Official approval from the ethics committee of the Republic of Slovenia was obtained for this study. After being informed about the research and potential risks, all patients giving written informed consent will undergo an orthopedic examination and those with a confirmed diagnosis of knee osteoarthritis that lasted more than 6 months will be included in the study. All participants were randomly divided into two groups. Participants in the first group receive single shot ACB and participants in the second group receive PRF therapy at the same point. Before starting all patients filled the Knee injury and osteoarthritis outcome(KOOS) form and estimated the maximal and minimal intensity of pain in the knee. They repeat self-assessment of pain, in the same manner, using 11 points numeric rating score(NRS) 1 month, 3, and six months after the blockade or PRF therapy. Measurement of maximum voluntary isometric contraction of the quadriceps muscle (MVIC), time up and go test(TUG), and 30s stand-up chair test are performed by a physiotherapist before a block of adductor canal on both legs,1 hour, 1 month, 3 months and 6 months after a block or PRF therapy.The adductor canal blockl is performed by the same trained anesthesiologist at the proximal part of the leg using 14 ml of Levobupivacaine and 100 mcg of Clonidine mixed in the same syringeAfterof the study participants filled the Knee injury and osteoarthritis outcome(KOOS) form once again.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of the Knee osteoarthritis confirmed by orthopedic examination
* K-L grades 3 and 4
* A sufficient level of education to understand study procedures
* Be able to communicate with site personnel
* Age >45 years

Exclusion Criteria :

* Any cardiovascular, hepatic, or renal conditions that would compromise participation, in the opinion of the investigator
* Severe neurologic conditions interfere with a knee condition
* Narcotic dependent (opioid intake of more than 3 months and more than 30 mg of daily oral morphine equivalents)
* Coexisting severe hematological disorder or deranged coagulation parameters
* Psychiatric illnesses
* Allergy to any of the drugs used in the study
* Infection or malignancy at the site of the block
* Any active systemic infection
* Implanted electronic devices like spinal cord stimulators, cardiac pacemakers or similar

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants included in this study were sent by family physicians to our Pain ambulance and all have already been diagnosed with knee osteoarthritis chronic pain. The diagnosis was confirmed by Orthopedist engaged in our study. Anesthesiologist decides if the patient is appropriate for the study.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline ,1 hour,1 month, 3 month and 6 months
  Change From Baseline in Maximal and minimal Pain on the 11-point Numeric rating score Pain Scale (NRS 0-11) ;Numeric 11-point rating score is widely accepted self-reported score for measurement of chronic and acute pain in researches.Possible scores range are between 0-free of pain and 10-the worst imaginable pain.
KOOS | Baseline ,1 hour,1 month, 3 month and 6 months
  The Knee injury and osteoarthritis outcome(KOOS) score change in percentage from baseline and 1 month following adductor canal block [ Time Frame: Baseline and 1 month following adductor canal block ] KOOS is valid,reliable outcome measure in patients with knee osteoarthritis. usually used following knee surgery.This method is recognised as useful also in other and nonsurgical knee treatment.Shortened version widely used in North America is western Ontario and McMaster Universities Index(WOMAC)

SECONDARY OUTCOMES:
Maximum voluntary isometric contraction of quadriceps muscle (MVIC) | Baseline ,1 hour,1 month, 3 month and 6 months
  Maximum voluntary isometric contraction of quadriceps muscle (MVIC) measured by handheld dynamometer ] This method is used to check impact of block on contraction of quadriceps muscle.
Timed up to go test (TUG) | Baseline ,1 hour,1 month, 3 month and 6 months
  Time that patient need to stand up from a standard height armchair,walk 3 meters,go back to the chair and takes a seat.Used to assess a patients balance,risk of falling and global mobility
Satisfaction of patient | Baseline ,1 hour,1 month, 3 month and 6 months
  We determine whether the patient is satisfied with the result of treatment by asking the following question: "what is the least amount of success that the treatment would have to achieve by the end of the study and/or treatment for the patient to conclude that the treatment was worth it and the patient is satisfied?" The patient is asked to describe the minimum goal to be satisfied with the treatment in her own words, such as: "50% reduction in pain, to go to the store without assistance, to use only one cane, to not wake up with pain, to perform regular housekeeping duties at home with minimal breaks, to walk a certain distance, or to play tennis". At the end of the study the patient indicates whether that goal was achieved with a "yes" or "no" answer.
Range of knee motion (ROM) | Baseline ,1 hour,1 month, 3 month and 6 months
  Passive knee joint ROM of extension and flexion was measured in the control and blocked leg in the supine position using a goniometer.
30 seconds stand up chair test (30 s SCT) | Baseline ,1 hour,1 month, 3 month and 6 months
  In the 30 s CST, number of times the participant rises from a chair in 30 s is counted.

CONTACTS AND LOCATIONS:
Overall Officials: Mensur Salihovic, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared with all other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the end of the study and the publishing results.
Access Criteria: The request needs to be addressed to the principal investigator. It should come from an official address or from a student or researcher personally.

REFERENCES:
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Ikeuchi M, Ushida T, Izumi M, Tani T. Percutaneous radiofrequency treatment for refractory anteromedial pain of osteoarthritic knees. Pain Med. 2011 Apr;12(4):546-51. doi: 10.1111/j.1526-4637.2011.01086.x. Epub 2011 Apr 4. PMID 21463469
- [Background] Salihovic M, Rijavec B, Muratagic A, Blagus R, Puh U. Effectiveness of Ultrasound-Guided Canal Adductor Blockade for Chronic Pain and Functioning in Knee Osteoarthritis: A Prospective Longitudinal Observational Study. Biomed Res Int. 2022 Jan 22;2022:5270662. doi: 10.1155/2022/5270662. eCollection 2022. PMID 35103237
- [Background] Burckett-St Laurant D, Peng P, Giron Arango L, Niazi AU, Chan VW, Agur A, Perlas A. The Nerves of the Adductor Canal and the Innervation of the Knee: An Anatomic Study. Reg Anesth Pain Med. 2016 May-Jun;41(3):321-7. doi: 10.1097/AAP.0000000000000389. PMID 27015545
- [Background] Akbas M, Luleci N, Dere K, Luleci E, Ozdemir U, Toman H. Efficacy of pulsed radiofrequency treatment on the saphenous nerve in patients with chronic knee pain. J Back Musculoskelet Rehabil. 2011;24(2):77-82. doi: 10.3233/BMR-2011-0277. PMID 21558611
- [Background] Carpenedo R, Al-Wardat M, Vizzolo L, Germani G, Chine E, Ridolfo S, Dauri M, Natoli S. Ultrasound-guided pulsed radiofrequency of the saphenous nerve for knee osteoarthritis pain: a pilot randomized trial. Pain Manag. 2022 Mar;12(2):181-193. doi: 10.2217/pmt-2021-0035. Epub 2021 Aug 25. PMID 34431329
- [Background] Zhang H, Wang B, He J, Du Z. Efficacy and safety of radiofrequency ablation for treatment of knee osteoarthritis: a meta-analysis of randomized controlled trials. J Int Med Res. 2021 Apr;49(4):3000605211006647. doi: 10.1177/03000605211006647. PMID 33887985
- [Background] Uematsu H, Osako S, Hakata S, Kabata D, Shintani A, Kawazoe D, Mizuno K, Fujino Y, Matsuda Y. A Double-Blind, Placebo-Controlled Study of Ultrasound-Guided Pulsed Radiofrequency Treatment of the Saphenous Nerve for Refractory Osteoarthritis-Associated Knee Pain. Pain Physician. 2021 Sep;24(6):E761-E769. PMID 34554694
- [Background] Gupta A, Huettner DP, Dukewich M. Comparative Effectiveness Review of Cooled Versus Pulsed Radiofrequency Ablation for the Treatment of Knee Osteoarthritis: A Systematic Review. Pain Physician. 2017 Mar;20(3):155-171. PMID 28339430
- [Result] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873